CLINICAL TRIAL: NCT06506747
Title: Clinical Evaluation of FastMap Navigated Photogrammetry for Assessing Implant Positions Compared to Standard Stereophotogrammetry
Brief Title: Navigated Photogrammetry Compared to Standard Stereophotogrammetry
Acronym: FSTMP
Status: Completed | Type: Observational
Sponsor: X-Nav Technologies, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DOC-002105
Record Dates: First submitted 2024-07-02; First posted 2024-07-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Doctor Efficiency; Dental Prosthesis Fit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- FastMap Navigated Photogrammetry: Following implant surgery, the patient will then receive a provisional that was manufactured using the data from FastMap Navigated Photogrammetry.
  Interventions: Device: Navigated Photogrammetry
- Standard Stereophotogrammetry: Following implant surgery, the patient will then receive a provisional that was manufactured using the data from Standard Stereophotogrammetry.
  Interventions: Device: Standard Photogrammetry

INTERVENTIONS:
Device: Navigated Photogrammetry — Navigated Photogrammetry shall be performed following implant surgery, rather than standard stereophotogrammetry. The patient will then receive a provisional that was manufactured using the data from FastMap Navigated Photogrammetry.
  Groups: FastMap Navigated Photogrammetry
Device: Standard Photogrammetry — The patient will receive the existing patient care protocol that includes anatomy information for the manufacturing of the provisional. Specifically, the patient will receive a preoperative IntraOral Scan (IOS) anatomy scan with IOS-compatible fiducials. Following implant surgery, the patient will receive a scan with a standard stereophotogrammetry device. Additionally, they will receive a post-op alignment IOS with IOS-compatible anatomy fiducials and IOS-compatible implant scan bodies. The patient will then receive a provisional that was manufactured using the data from the standard stereophotogrammetry device.
  Groups: Standard Stereophotogrammetry

SUMMARY:
The purpose of this study is to compare the clinical outcome of Navigated Photogrammetry to standard stereophotogrammetry techniques in digital dentistry for the following two parameters:

* The amount of time needed to prepare the provisional digital files for use in the lab, measured in direct doctor interaction time.
* Suitability of delivered provisional occlusion.

Participants will receive either a provisional manufactured by the output of Navigated Photogrammetry, or a provisional manufactured by the output of standard stereophotogrammetry.

DETAILED DESCRIPTION:
Prior to implant surgery, a patient treatment plan is developed using a cone-beam computed tomography (CBCT), Intra Oral Scan (IOS), or digitized analog records. These records are loaded into a computer-aided design (CAD) program. The individual planning files are all related to one another in one coordinate system. This plan can be used to produce provisional restorations via computer-aided manufacturing (CAM). These files can also be used to implement the plan during surgery using either static guides or dynamic navigation.

Following implant surgery, the final placed implant locations will inherently have some deviation from the plan. It is important for the dentist to understand the physical location of the placed implants to achieve passive fit. In implant dentistry, a "passive fit" refers to the precise alignment and seating of prosthetic components onto dental implants without any internal stress or strain. Achieving a passive fit is crucial for the long-term success and stability of the dental prosthesis.

A potential method to obtain the final implant locations is stereophotogrammetry. Navigated Photogrammetry (NPG) is a new form of stereophotogrammetry which is inherently capable of relating the placed implants to the patient's anatomy using the registration of the Dynamic Surgical Navigation System (DSNS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring dental implant reconstruction who would undergo implant surgery with or without participation in the study.
* The patient must need at least four implants placed in one or both jaws of the maxilla or mandible.
* All patients must undergo informed consent and willingly read, understand, and accept the risks and benefits associated with the study.
* Willingness to participate for the duration of the study of at least six months follow-up
* Is healthy enough to undergo implant surgery. i.e. patient is classified by the American Society of Anesthesiology Scale (ASA) physical status classification status as ASA 1, 2 or 3.
* Ample bone to fully accommodate the implants without impinging on vital structures.

Exclusion Criteria:

* Patients who are not candidates for implant placement.
* Children and adolescents under 21 years of age.
* Refusal to sign informed consent.
* Less than four implants need to be restored.
* Severely immunocompromised patients
* Patients undergoing chemotherapy
* Pregnant females.
* Classified by the ASA physical status classification status as ASA > 3,
* Patient at high risk for medication induced osteonecrosis of the jaw or any other medical condition that would preclude implant placement,
* Any systemic or local disease or condition that would compromise post healing and /or osseointegration.
* Need for systemic corticosteroids or any other medication that would compromise postoperative healing and / or osseointegration.
* Current alcohol or drug abuse.
* Inability or willingness to return for follow-up visits for the period of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be current patients of the investigators who are already intended to undergo implant placement surgery. Participants who willingly accepted the risks and benefits associated with placement of dental implants and stereophotogrammetry in the private practice of the investigators will be considered for inclusion in the study. Those patients deemed ineligible or who chose not to participate in the research study will be treated using conventional techniques.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Provisional prosthesis fit | at provisional placement completion, approximately 2 weeks
  The passive fit of the provisional prosthesis onto the implants as well as occlusal fit with the opposing jaw.
Clinician interaction time | at provisional placement completion, approximately 2 weeks
  The amount of time needed to prepare each type of provisional digital files for use in the lab, measured in direct doctor interaction time.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Center For Oral and Maxillofacial Surgery and For Cosmetic Surgery, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pozzi A, Agliardi E, Lio F, Nagy K, Nardi A, Arcuri L. Accuracy of intraoral optical scan versus stereophotogrammetry for complete-arch digital implant impression: An in vitro study. J Prosthodont Res. 2024 Jan 16;68(1):172-180. doi: 10.2186/jpr.JPR_D_22_00251. Epub 2023 Aug 11. PMID 37574278
- [Background] Orejas-Perez J, Gimenez-Gonzalez B, Ortiz-Collado I, Thuissard IJ, Santamaria-Laorden A. In Vivo Complete-Arch Implant Digital Impressions: Comparison of the Precision of Three Optical Impression Systems. Int J Environ Res Public Health. 2022 Apr 3;19(7):4300. doi: 10.3390/ijerph19074300. PMID 35409985
- [Background] Revilla-Leon M, Att W, Ozcan M, Rubenstein J. Comparison of conventional, photogrammetry, and intraoral scanning accuracy of complete-arch implant impression procedures evaluated with a coordinate measuring machine. J Prosthet Dent. 2021 Mar;125(3):470-478. doi: 10.1016/j.prosdent.2020.03.005. Epub 2020 May 6. PMID 32386912
- [Background] Revilla-Leon M, Rubenstein J, Methani MM, Piedra-Cascon W, Ozcan M, Att W. Trueness and precision of complete-arch photogrammetry implant scanning assessed with a coordinate-measuring machine. J Prosthet Dent. 2023 Jan;129(1):160-165. doi: 10.1016/j.prosdent.2021.05.019. Epub 2021 Jun 18. PMID 34154820
- [Background] Tohme H, Lawand G, Chmielewska M, Makhzoume J. Comparison between stereophotogrammetric, digital, and conventional impression techniques in implant-supported fixed complete arch prostheses: An in vitro study. J Prosthet Dent. 2023 Feb;129(2):354-362. doi: 10.1016/j.prosdent.2021.05.006. Epub 2021 Jun 8. PMID 34112521
- [Background] Manzella C, Bignardi C, Burello V, Carossa S, Schierano G. Method to improve passive fit of frameworks on implant-supported prostheses: An in vitro study. J Prosthet Dent. 2016 Jul;116(1):52-8. doi: 10.1016/j.prosdent.2016.01.006. Epub 2016 Mar 2. PMID 26944406
- [Background] Jemt T, Hjalmarsson L. In vitro measurements of precision of fit of implant-supported frameworks. A comparison between "virtual" and "physical" assessments of fit using two different techniques of measurements. Clin Implant Dent Relat Res. 2012 May;14 Suppl 1:e175-82. doi: 10.1111/j.1708-8208.2011.00416.x. Epub 2011 Dec 15. PMID 22171700
- [Background] Schwarz MS. Mechanical complications of dental implants. Clin Oral Implants Res. 2000;11 Suppl 1:156-8. doi: 10.1034/j.1600-0501.2000.011s1156.x. PMID 11168264
- See also: Accuracy (trueness and precision) of measurement methods and results-Part 1: General principles and definitions — https://www.iso.org/obp/ui/es/#iso:std:iso:5725:-1:en